CLINICAL TRIAL: NCT06002009
Title: SupraScapular Cuff Study: Assessing the Effects of Size and Type of Rotator Cuff Tear on Suprascapular Nerve Function
Acronym: SSCuFF
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3103
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Orthopedic Disorder
Keywords: Rotator cuff tear; Suprascapular nerve function
MeSH Terms: conditions — Musculoskeletal Diseases; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MRI — MRI of shoulder
Other: Nerve conduction study — Nerve conduction study

SUMMARY:
The primary objective of the study is to determine in adult patients with a rotator cuff tear, what size and pattern of rotator cuff tear would result in damage to the suprascapular nerve.

The secondary objectives are

1. To determine if an injured suprascapular nerve can recover if the rotator cuff tear is surgically repaired.
2. To determine if there is a limit of retraction before the suprascapular nerve is irreversibly damaged.
3. To determine factors that are protective against SSN injury.
4. Can the patient data gathered be used to optimise operative procedures.

ELIGIBILITY:
Inclusion Criteria:

• All patients age ≥18 years presenting to a UHNM shoulder clinic with a confirmed diagnosis of a rotator cuff tear (affecting one or both shoulders).

Exclusion Criteria:

* Bony pathology (such as significant shoulder arthritis that would exclude isolated rotator cuff repair)
* Grossly abnormal shoulder anatomy
* Motor Neurone Disease
* Cervical cord disease affecting the SSN nerve roots
* Patients unable to undergo MRI scan
* Previous surgery at the affected glenohumeral joint
* Patients unable to tolerate NCS
* Acute fracture affecting the glenohumeral joint
* Recent glenohumeral joint dislocation (past 12 months)
* Patients unable or unwilling to give full informed consent
* Patients unable or unwilling to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the University Hospitals of North Midlands outpatient clinic
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Assess suprascapular nerve funaction | 36 months
  MRI scan to quantify size of rotator cuff tear, compared with Nerve Conduction Studies (NCS) to assess suprascapular nerve function.

SECONDARY OUTCOMES:
Shoulder scores | 36 months
  Compare functional shoulder scores to the degree of nerve injury and muscle degeneration over a 24-month period post-injury. Scores to include active range of movement (ROM) measurements; and the collection of validated shoulder outcome scores (DASH, OSS, & Constant score).
Nerve recovery | 24 months
  Functional assessment of nerve recovery at 24 months post-injury for surgically repaired rotator cuff tears.
Machine learning | 24 months
  Use of machine learning to investigate data set for optimum parameters or predictors
Nerve conduction studies | 12 months
  Repeat Nerve Conduction Study investigations at 12 months post injury for all surgically managed participants and non-surgical patients to assess suprascapular nerve function

CONTACTS AND LOCATIONS:
Overall Officials: Damian McClelland, Principal Investigator — University Hospital of North Midlands NHS Trust
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No